CLINICAL TRIAL: NCT04730466
Title: Validation of Cognitive Rehabilitation as a Balance Rehabilitation Strategy in Patients With Parkinson's Disease: Study Protocol for a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation as a Balance Rehabilitation Strategy in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Hospital Beata María Ana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Balanc-EP
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Balance; Information Processing Speed
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study will be a parallel, randomized and controlled experimental study. The patients included in the sample will be randomly distributed into two groups: Cognitive rehabilitation (experimental) and No therapy (control). The randomization of the sample will be carried out through the website: http://www.randomization.com/.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuropsychological rehabilitation (Experimental): In the experimental group, patients will receive a 12-session neuropsychological rehabilitation protocol that will be carried out over four weeks (3 weekly sessions). The protocol and the number of sessions has been designed by neuropsychologists following the Díez-Cirarda et al. recommendations
  Interventions: Other: Neuropsychological rehabilitation
- Control (No Intervention): The control group will not receive any therapy. The participants will be simply evaluated at the same time as the experimental group

INTERVENTIONS:
Other: Neuropsychological rehabilitation — The intervention can be carried out in the research unit or in the Parkinson's association. Each session will consist of a series of cognitive stimulation tasks aimed at improving attention, perception and processing speed. These tasks will be applied through the NeuronUp cognitive neurorehabilitation platform to achieve maximum homogeneity and objectivity in their application. The program is programmed and is identical for all patients. Performing tasks through the platform allows us to objectively record the performance of each patient in all tasks.
  Arms: Neuropsychological rehabilitation

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder. PD is characterized by motor symptoms, such as bradykinesia, tremor, and rigidity. Although balance impairment is characteristic of advanced stages, it can be present with less intensity since the beginning of the disease. Approximately 60% of PD patients fall once a year and 40% recurrently These falls may be correlated with the inability to achieve compensatory movements to regain balance when their center of gravity tends to swing outside their range of stability, which is reduced in this disease. On the other hand, cognitive symptoms affect up to 20% of patients with PD in early stages and can even precede the onset of motor symptoms. There are cognitive requirements for balance and can be challenged when attention is diverted or reduced, linking a worse balance and a higher probability of falls with a slower cognitive processing speed and attentional problems. Cognitive rehabilitation of attention and processing speed can lead to an improvement in postural stability in patients with Parkinson's. The investigators present a parallel and controlled Randomized Clinical Trial (RCT) to assess the impact on balance of a protocol based on cognitive rehabilitation focused on sustained attention through the NeuronUP platform (Neuronup SI, La Rioja, España) in patients with PD. This therapy opens the possibility of new rehabilitation strategies for prevention of falls in PD, reducing morbidity and saving costs to the health system.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder. This disease is characterized by motor symptoms, such as bradykinesia, tremor, and rigidity. Non-motor symptoms such as cognitive impairment, anosmia, sleep disorders, or depression are also part of the disease, and although their prevalence is very high, non-motor symptomsare often underdiagnosed.

One of the cognitive characteristics in PD is the slowness in the processing of information, which includes deficits in processing speed and attention, cognitive inflexibility, and forgetfulness. These symptoms may appear from the initial stages of the disease.

Approximately 60% of PD patients fall once a year and 40% do so regularly. These falls may be correlated with the inability to achieve compensatory movements to regain balance when their center of gravity generally oscillates outside their limits of stability (LOS), which is reduced in this disease. Some authors point out that reaction times and processing speed may be a marker of postural instability since a reduced speed is associated with difficulty in making turns. This is in line with Pantall's findings, indicating that cognitive function and postural control normally progressively worsen with disease progression.

The relationship between cognitive impairment and postural instability in PD patients may be specific for tasks that assess the dorsolateral prefrontal cortex and its frontal-subcortical connections. The main cognitive functions whose affectation would influence a worse balance and gait performance would be attention and executive functions. Varalta et al specified that balance is related to executive functions and attention, while functional mobility is more related to cognitive impairment, verbal fluency, and attentional capacity.

Some authors point out that within the executive functions the component with the greatest weight in this relationship would be the inhibitory control. Dual-task performance has also been established as a good indicator of falls in patients with early-stage PD and no previous history of falls. The studies that carried out a one and a half years follow-up of the participants concluded that the deterioration of executive functions acts as a predictor of future falls in patients with PD.

Cognitive rehabilitation through neurorehabilitation platforms and neuropsychological rehabilitation in patients with Parkinson's disease has shown to be effective in improving processing speed, attention, and executive functions.

Although the relationship between cognitive deficits and postural stability seems to be demonstrated, the investigators have not found studies that, through cognitive rehabilitation, seek a stability improvement.

The investigators working hypothesis is that the group that receives rehabilitation of the speed of information processing and sustained attention will improve their postural stability compared to the group that does not undergo any therapy.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (diagnosed according to the UK Parkinson´s Disease Society Brain Bank criteria).
* Stage <III Hoehn-Yahr with no obvious motor fluctuations.

Exclusion Criteria:

* Visual-perceptual difficulties.
* Peripheral sensory disturbances due to polyneuropathy.
* Cerebellar alterations.
* Severe cognitive impairment (MoCA <24).
* Moderate or severe active depression (BDI> 14).
* Dependence (mRS> 3).
* Dopaminergic medication changes in the last 30 days.
* Structural changes MRI Severe comorbidity (cancer, severe COPD ...).
* Atypicality data for idiopathic PD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Change in Timed stand up and go test score | From Baseline at 5 weeks
  The timed "Up and Go" test measures, in seconds, the time it takes a person to get up from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down again.
Change in Berg Balance scale score | From Baseline at 5 weeks
  Consists of 14 items scored on an ordinal scale of 0 to 4 for a total of 56 points (a higher score indicates lower fall risk). Scale is designed to measure changes in functional standing balance over time. This scale measures the balance skills observed during tasks that involve sitting, standing, and changing positions.
Change in Stability limits test: The Biodex Stability Limits (LOS) score | From Baseline at 5 weeks
  This test is a challenge for the patient when it comes to moving and exercising control over gravity supported on a base. During each test the patient must change their weight to move the cursor from the center of the target to a new point that will flash on the screen and that will change as fast as the slightest movement or deviation is noticed. This same process will be repeated until another nine objectives are achieved. The test dependent variables provided by the machine are the time (seconds) it takes for the subject to complete the test and the directional control value which is the proportion of the distance travelled by the cursor from the center to each target (based on that 100% is a straight line from the center to the intended target). This means that the greater the distance travelled by the subject, the worse their stability.
Change in Fall risk test score | From Baseline at 5 weeks
  During the test, the patient undergoes three attempts of 20 seconds each, beginning with an initial platform mobility setting of 6 and ending with a platform setting of 2 (from least to most mobile), with rest periods ten seconds between each test. The patient stands with feet shoulder-width apart on the midline of the board. At the end of the index test it is calculated according to the degree of instability of the patient with each configuration. Own normative data are applied.
Finger tapping (FT) | Baseline
  The FT task has been used as a measure of motor function. In this task, following the Strauss application guidelines, participants are instructed to press the space bar on the keyboard as quickly as possible and repeatedly with the index finger. Five 10-second attempts are made with the dominant hand. The average time between two consecutive hits in the five trials is the dependent variable.
Finger tapping (FT) | At 5 weeks from baseline
  The FT task has been used as a measure of motor function. In this task, following the Strauss application guidelines, participants are instructed to press the space bar on the keyboard as quickly as possible and repeatedly with the index finger. Five 10-second attempts are made with the dominant hand. The average time between two consecutive hits in the five trials is the dependent variable.
Simple reaction time (SRT) | Baseline
  This task is used as a measure of simple perception and sustained alertness. Participants are instructed to press the left mouse button as fast as possible when the stimulus "+" appears in the center of the screen with a size of 2 cm x 2 cm. The order of appearance is constant for all participants. The task consists of 50 trials that lasted 2-3 minutes.The average time between the stimulus and the response is the dependent variable.
Simple reaction time (SRT) | At 5 weeks from baseline
  This task is used as a measure of simple perception and sustained alertness. Participants are instructed to press the left mouse button as fast as possible when the stimulus "+" appears in the center of the screen with a size of 2 cm x 2 cm. The order of appearance is constant for all participants. The task consists of 50 trials that lasted 2-3 minutes.The average time between the stimulus and the response is the dependent variable.
Simple task of attention to sustained response time (SRT-SART) | Baseline
  This task helps us to measure the inhibitory response strategy. The participants have to press the left mouse button when the stimulus (digits 1-9) appears in the center of the screen and inhibit the response when it appears as the number "3". The task consists of 168 Go trials and 21 No / Go ; the average duration is 4 minutes. The stimuli vary in size between 12 mm and 29 mm.The average time between the stimulus and the response is the dependent variable.
Simple task of attention to sustained response time (SRT-SART) | At 5 weeks from baseline
  This task helps us to measure the inhibitory response strategy. The participants have to press the left mouse button when the stimulus (digits 1-9) appears in the center of the screen and inhibit the response when it appears as the number "3". The task consists of 168 Go trials and 21 No / Go ; the average duration is 4 minutes. The stimuli vary in size between 12 mm and 29 mm.The average time between the stimulus and the response is the dependent variable.
Choice reaction time (CRT) | Baseline
  This task was used as a measure of visual perception decision time and is related to the same processes involved in the SRT plus the processing of the uncertainty about which of the stimuli will appear to the continuation, that is, decisional processing. Participants have to press the left mouse button when a square appears in the center of the screen (4 cm x 4 cm) or press the right button when a circle appears. The task consists of 80 tests with a duration of approximately 3 minutes.The average time between the stimulus and the response is the dependent variable.
Choice reaction time (CRT) | At 5 weeks from baseline
  This task was used as a measure of visual perception decision time and is related to the same processes involved in the SRT plus the processing of the uncertainty about which of the stimuli will appear to the continuation, that is, decisional processing. Participants have to press the left mouse button when a square appears in the center of the screen (4 cm x 4 cm) or press the right button when a circle appears. The task consists of 80 tests with a duration of approximately 3 minutes.The average time between the stimulus and the response is the dependent variable.
Choice-search reaction time (CRT-Search) | Baseline
  This task helps us to measure visual search. Participants have to press the left mouse button when a "Z" appears in a 6-letter sequence or press the right button when it does not appear. Stimuli are classified according to two dimensions: presence/absence of "Z". The task consists of 128 trials that lasted between 5 and 8 minutes. The average time between the stimulus and the response is the dependent variable.
Choice-search reaction time (CRT-Search) | At 5 weeks from baseline
  This task helps us to measure visual search. Participants have to press the left mouse button when a "Z" appears in a 6-letter sequence or press the right button when it does not appear. Stimuli are classified according to two dimensions: presence/absence of "Z". The task consists of 128 trials that lasted between 5 and 8 minutes. The average time between the stimulus and the response is the dependent variable.
Stroop test | Baseline
  The standardized version applied consists of three DIN-A4 size sheets. Each of which contains 100 elements distributed in five columns of 20 elements. On the first sheet (Stroop-P), the words 'RED', 'GREEN' and 'BLUE' appear, arranged at random and printed in black ink, and the examinee must read them. On the second sheet (Stroop C), all the elements have the same shape ('XXXX') but printed in blue, green, or red ink, and the examinee must say out loud what the color of each one is. On the third sheet (Stroop PC), the first sheet words appear printed in the colors of the second, and the examinee must name the color of the ink with which the word is printed, ignoring the meaning. For each of the sheets, the subject has 45 seconds to say as many items as possible. The number of items and errors are counted for each of the conditions
Stroop test | At 5 weeks from baseline
  The standardized version applied consists of three DIN-A4 size sheets. Each of which contains 100 elements distributed in five columns of 20 elements. On the first sheet (Stroop-P), the words 'RED', 'GREEN' and 'BLUE' appear, arranged at random and printed in black ink, and the examinee must read them. On the second sheet (Stroop C), all the elements have the same shape ('XXXX') but printed in blue, green, or red ink, and the examinee must say out loud what the color of each one is. On the third sheet (Stroop PC), the first sheet words appear printed in the colors of the second, and the examinee must name the color of the ink with which the word is printed, ignoring the meaning. For each of the sheets, the subject has 45 seconds to say as many items as possible. The number of items and errors are counted for each of the conditions
The Bells Test | Baseline
  This task is a distractor instrument that requires a horizontal visual examination on a sheet of A4 size. The target stimuli are bell figures and are located in a pseudo-random way, organized in seven columns containing five bells each one. The columns are positioned on the sheet as follows: three on the left side, one in the middle, and three on the right side of the paper.The task is completed when the subject stops her activity. The time of completion of the test, the number of hits and omissions is counted.
The Bells Test | At 5 weeks from baseline
  This task is a distractor instrument that requires a horizontal visual examination on a sheet of A4 size. The target stimuli are bell figures and are located in a pseudo-random way, organized in seven columns containing five bells each one. The columns are positioned on the sheet as follows: three on the left side, one in the middle, and three on the right side of the paper. The task is completed when the subject stops her activity. The time of completion of the test, the number of hits and omissions is counted.
Trail Making Test | Baseline
  It is a measure of combined speed for attention, sequencing, visual and mental searching, as well as motor function. It is made up of two parts: A and B. While part A fundamentally requires visual-perceptual skills, part B requires working memory functioning, as well as skills to change tasks. The task ends when the subject completes the test. The examiner corrects errors during the task, taking the subject to the previous item. The task completion time is measured.
Trail Making Test | At 5 weeks from baseline
  It is a measure of combined speed for attention, sequencing, visual and mental searching, as well as motor function. It is made up of two parts: A and B. While part A fundamentally requires visual-perceptual skills, part B requires working memory functioning, as well as skills to change tasks. The task ends when the subject completes the test. The examiner corrects errors during the task, taking the subject to the previous item. The task completion time is measured
Digit Span | Baseline
  The test is part of the WAIS-III. The examiner reads aloud a series of digits at a rate of one per second and the examinee must repeat this series thereafter in the same order as it was presented (direct digits) or in the reverse order (reverse digits). The test begins with a two-digit series. In each test two series of equal length are read and, if the examinee correctly repeats at least one of the two, the next test is continued in which the series has one digit more than the previous ones. The test ends when the examinee does not pass two series of the same duration. Each of the said series of digits is scored with a point. The sum of the points in each condition (direct and inverse), the sum of both scores and the maximum number of digits said in a series, will be the dependent variables.
Digit Span | At 5 weeks from baseline
  The test is part of the WAIS-III. The examiner reads aloud a series of digits at a rate of one per second and the examinee must repeat this series thereafter in the same order as it was presented (direct digits) or in the reverse order (reverse digits). The test begins with a two-digit series. In each test two series of equal length are read and, if the examinee correctly repeats at least one of the two, the next test is continued in which the series has one digit more than the previous ones. The test ends when the examinee does not pass two series of the same duration. Each of the said series of digits is scored with a point. The sum of the points in each condition (direct and inverse), the sum of both scores and the maximum number of digits said in a series, will be the dependent variables
FAS Word Fluency | Baseline
  In this task, the examinee is asked to produce the most number of words belonging to a restricted category within a limited time (60 seconds). The assessment of verbal fluency is divided into two tests: 1) semantic verbal fluency: where the subject is asked to name all the elements within a given semantic category (animals), and 2) phonological verbal fluency: where the subject has to name all the elements that start with a particular letter (F, A, and S), not being able to say proper names and words derived from others previously said.The number of correct words, the number of perseverations, proper names and derived words in each of the conditions will be accounted
FAS Word Fluency | At 5 weeks from baseline
  In this task, the examinee is asked to produce the most number of words belonging to a restricted category within a limited time (60 seconds). The assessment of verbal fluency is divided into two tests: 1) semantic verbal fluency: where the subject is asked to name all the elements within a given semantic category (animals), and 2) phonological verbal fluency: where the subject has to name all the elements that start with a particular letter (F, A, and S), not being able to say proper names and words derived from others previously said. The number of correct words, the number of perseverations, proper names and derived words in each of the conditions will be accounted
Processing Speed-Digit Symbol Coding | Baseline
  It is a subtest that is part of the Wechsler Adult Intelligence Scale (WAIS-III). It consists of a sheet in which 9 different aligned symbols are presented in the upper part, to which a consecutive number from 1 to 9 has been assigned. In the lower part, numbers from 1 to 9 appear in random order, and below each one of them a blank space in which the examinee must draw the corresponding symbol. The duration of the task is two minutes and the number of hits and errors are quantified
Processing Speed-Digit Symbol Coding | At 5 weeks from baseline
  It is a subtest that is part of the Wechsler Adult Intelligence Scale (WAIS-III). It consists of a sheet in which 9 different aligned symbols are presented in the upper part, to which a consecutive number from 1 to 9 has been assigned. In the lower part, numbers from 1 to 9 appear in random order, and below each one of them a blank space in which the examinee must draw the corresponding symbol. The duration of the task is two minutes and the number of hits and errors are quantified.
Processing Speed-Symbol Search | Baseline
  It is a subtest included in the Wechsler Adult Intelligence Scale (WAIS-III). It consists of several plates in which two symbols are presented and next to them, another set of 5. The person must decide if any of the first two symbols appear in the second group, marking yes or no in the corresponding place. The duration of the task is two minutes and the number of hits and errors are quantified
Processing Speed-Symbol Search | At 5 weeks from baseline
  It is a subtest included in the Wechsler Adult Intelligence Scale (WAIS-III). It consists of several plates in which two symbols are presented and next to them, another set of 5. The person must decide if any of the first two symbols appear in the second group, marking yes or no in the corresponding place. The duration of the task is two minutes and the number of hits and errors are quantified

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire 39 | Baseline
  It is a specific questionnaire for evaluating the health status of Parkinson's patients. It is a multidimensional scale in which the subjects have to affirm one among five answers ordered in categories according to how frequent, due to Parkinson's disease, the patients have experienced the problem defined by each item. The items are grouped into 8 scales and are scored by expressing the sum of the scores for each item as a percentage that can be between 0 and 100%. Higher scores indicate poorer quality of life
Parkinson's Disease Questionnaire 39 | At 5 weeks from baseline
  It is a specific questionnaire for evaluating the health status of Parkinson's patients. It is a multidimensional scale in which the subjects have to affirm one among five answers ordered in categories according to how frequent, due to Parkinson's disease, the patients have experienced the problem defined by each item. The items are grouped into 8 scales and are scored by expressing the sum of the scores for each item as a percentage that can be between 0 and 100%. Higher scores indicate poorer quality of life
Resting EEG | Baseline
  The spectral entropy correlation, the coherence and interhemispheric divergence will be analyzed in a 64-channel resting EEG
Resting EEG | At 5 weeks from baseline
  The spectral entropy correlation, the coherence and interhemispheric divergence will be analyzed in a 64-channel resting EEG
Tapping EEG | Baseline
  A 64-channel EEG recording will be made while pressing for 30 seconds. The registration will be independent for each hand, starting with the dominant one. The spectral entropy correlation, the coherence and interhemispheric divergence will be analyzed in a 64-channel tapping EEG
Tapping EEG | At 5 weeks from baseline
  A 64-channel EEG recording will be made while pressing for 30 seconds. The registration will be independent for each hand, starting with the dominant one. The spectral entropy correlation, the coherence and interhemispheric divergence will be analyzed in a 64-channel tapping EEG

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Romero Muñoz, MD PhD, Principal Investigator — Universidad Francisco de Vitoria, Facultad de Ciencias Experimentales
Locations (1):
- Hospital Beata María Ana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be available to other researchers under request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months at the end of the study
Access Criteria: Individual anonymized participant data will be available to other researchers under request

REFERENCES:
- [Background] Shipley BA, Deary IJ, Tan J, Christie G, Starr JM. Efficiency of temporal order discrimination as an indicator of bradyphrenia in Parkinson's disease: the inspection time loop task. Neuropsychologia. 2002;40(8):1488-93. doi: 10.1016/s0028-3932(01)00195-6. PMID 11931953
- [Background] Dona F, Aquino CC, Gazzola JM, Borges V, Silva SM, Gananca FF, Caovilla HH, Ferraz HB. Changes in postural control in patients with Parkinson's disease: a posturographic study. Physiotherapy. 2016 Sep;102(3):272-9. doi: 10.1016/j.physio.2015.08.009. Epub 2015 Oct 3. PMID 26582134
- [Background] Allcock LM, Rowan EN, Steen IN, Wesnes K, Kenny RA, Burn DJ. Impaired attention predicts falling in Parkinson's disease. Parkinsonism Relat Disord. 2009 Feb;15(2):110-5. doi: 10.1016/j.parkreldis.2008.03.010. Epub 2008 May 19. PMID 18487069
- [Background] Pal G, O'Keefe J, Robertson-Dick E, Bernard B, Anderson S, Hall D. Global cognitive function and processing speed are associated with gait and balance dysfunction in Parkinson's disease. J Neuroeng Rehabil. 2016 Oct 28;13(1):94. doi: 10.1186/s12984-016-0205-y. PMID 27793167
- [Background] Varalta V, Picelli A, Fonte C, Amato S, Melotti C, Zatezalo V, Saltuari L, Smania N. Relationship between Cognitive Performance and Motor Dysfunction in Patients with Parkinson's Disease: A Pilot Cross-Sectional Study. Biomed Res Int. 2015;2015:365959. doi: 10.1155/2015/365959. Epub 2015 Mar 31. PMID 25918713
- [Background] Diez-Cirarda M, Ibarretxe-Bilbao N, Pena J, Ojeda N. Neurorehabilitation in Parkinson's Disease: A Critical Review of Cognitive Rehabilitation Effects on Cognition and Brain. Neural Plast. 2018 May 6;2018:2651918. doi: 10.1155/2018/2651918. eCollection 2018. PMID 29853840
- [Background] Stegemoller EL, Wilson JP, Hazamy A, Shelley MC, Okun MS, Altmann LJ, Hass CJ. Associations between cognitive and gait performance during single- and dual-task walking in people with Parkinson disease. Phys Ther. 2014 Jun;94(6):757-66. doi: 10.2522/ptj.20130251. Epub 2014 Feb 20. PMID 24557652
- [Background] Strauss, E.; Sherman, E.M.S.; Spreen, O.; Spreen, O. A compendium of neuropsychological tests: administration, norms, and commentary; 3rd ed.; Oxford University Press: Oxford ; New York, 2006; ISBN 978-0-19-515957-8.
- [Background] Lubrini G, Rios Lago M, Perianez JA, Tallon Barranco A, De Dios C, Fernandez-Fournier M, Diez Tejedor E, Frank Garcia A. The contribution of depressive symptoms to slowness of information processing in relapsing remitting multiple sclerosis. Mult Scler. 2016 Oct;22(12):1607-1615. doi: 10.1177/1352458516661047. PMID 27742916